CLINICAL TRIAL: NCT03919214
Title: Hypertension Management in Cancer Patients: Bringing PCPs "Back" Into Cancer Care
Brief Title: Hypertension Management in Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Initially suspended due to Covid-19. After much consideration, it was determined that we do not have the bandwidth to resume recruitment or any activities for this project.
Sponsor: Duke University (Other)
Collaborators: Duke Institute for Health Innovation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00102260
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Blood Pressure; Hypertension; Cancer; Cancer, Breast; Cancer of Prostate; CLL; Hematopoietic Malignancy
MeSH Terms: conditions — Hypertension; Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QardioArm and Messaging System (Other): Participants will self-monitor their blood pressure using the Qardio Bluetooth device and obtain 3 separate blood pressure measurements per week (2 morning, 1 evening) for 12 weeks. An automated messaging system for blood pressure management will be triggered by a weekly average systolic blood pressure >140 mm Hg or diastolic blood pressure >90 mm Hg. This automated message will be sent to the participant's primary care provider, with copies to the participant and the primary medical oncologist.
  Interventions: Other: Automated Messaging

INTERVENTIONS:
Other: Automated Messaging — This is a 12-week prospective study with two phases. Participants will use the QardioArm device to obtain 3 separate blood pressure measurements per week (2 morning, 1 evening). The QardioArm device will only be used as a tool to gather data. In Phase 1 (Weeks 1-4), participants will self-monitor their blood pressure using the Qardio Bluetooth device. In Phase 2 (Weeks 5-12), we will implement the auto-messaging system triggered by a weekly average systolic blood pressure >140 mm Hg or diastolic blood pressure >90 mm Hg.
  Other Names: QardioArm Blood Pressure Measurements and Automated Messaging

SUMMARY:
The investigators propose to leverage new technology using the Qardio app for iPhone and Android devices to automatically upload blood pressures, using a well-validated blue tooth blood pressure monitor (QardioArm), directly into the Duke electronic health record system (EPIC). Further, the investigators propose to develop an automated EHR (electronic health record) messaging system utilizing the home blood pressures that will be sent to the participant's PCP, with copies to the participant and the primary oncologist. This is a 12-week prospective non-randomized implementation study. 40 patients who are 18-74 years old who fall under the following criteria will be screened: 10 women with Stage 1-III breast cancer who are receiving either an anthracycleine of antiHER2 therapy, 10 men with prostate cancer on ADT, 10 individuals with CLL on ibrutinib therapy, and 10 individuals who are hematopoietic stem cell transplantation (HSCT) survivors. In Phase 1 (Weeks 1-4) of the study, participants will self-monitor their blood pressure using the QardioArm wireless upper arm blood pressure monitor 3 times per week. In Phase 2 (Weeks 5-12), the investigators will implement the auto-messaging system triggered by an abnormal weekly average systolic or diastolic blood pressure. The investigators will adapt the conceptual framework of Muldoon and colleagues whereby home blood pressure monitoring is combined with office blood pressures to optimize data for the primary care provider's clinical decision making. {Participants will be asked to complete a paper survey, upon enrollment, that will include life chaos and medication adherence questions. There will also be an end-of-study feedback survey (usability and acceptability questions through REDCap) for both the participants and their primary care providers. This is an implementation study with a descriptive analysis. The data generated from the study will be used in future studies, including testing of different interventions aimed at optimizing blood pressure control among patients on active cancer therapy. This study presents no greater than minimal risk to the subjects and adverse events are not anticipated.

DETAILED DESCRIPTION:
This is a 12-week prospective study with two phases. In Phase 1 (Weeks 1-4), participants will self-monitor their blood pressure using the Qardio bluetooth device. In Phase 2 (Weeks 5-12), the investigators will implement the auto-messaging system triggered by a weekly average systolic blood pressure >140 mm Hg or diastolic pressure >90 mm Hg. As per the recommendation of the ACC/AHA, the target blood pressure for patients with Stage A (at risk for heart failure) is systolic <130 / diastolic <80. This guideline is also consistent with the ACC/AHA blood pressure guideline for patients at risk for myocardial infarction. For this pilot study, our target blood pressure in messaging to Duke primary care providers will be <140 mm Hg and <90 mm Hg. For this study, the investigators will adapt the conceptual framework of Muldoon and colleagues whereby home blood pressure monitoring is combined with office blood pressures to optimize data for the PCP's clinical decision-making.

The investigators will use the QardioArm wireless upper arm blood pressure monitor. The investigators opted to use this device because it is validated, and has been approved to be integrated into the Duke EHR system. This QardioArm monitor is compatible with both iPhone and Android devices, which will provide an efficient method of transferring Bluetooth data to Epic. Within Epic, the home blood pressures will be uploaded directly from a smartphone to REVIEW FLOWSHEETS, MYCHART HEALTKIT TRACKER.

Participants will use the QardioArm device to obtain 3 separate blood pressure measurements per week (2 morning, 1 evening). The 2 morning blood pressure measurements will be taken between 5-11am before any caffeine intake or exercise. The evening blood pressure measurement will be taken between 4-12pm. During Phase 1, the investigators will review the individual and weekly average blood pressures and identify values that appear to be in error. This review will be used to refine the system and further train the participants on home blood pressure measurements if needed. Also during this phase, the investigators will develop the Blood Pressure Management Clinical Pathway for Patients and Survivors, based upon the ACC/AHA blood pressure guidelines and the ACC/AHA guidelines for prevention of cardiotoxicity. Lastly, in this phase, the investigators will develop the primary care provider messages to be implemented in Phase 2. These short messages will alert the Duke primary care provider that an abnormal weekly average blood pressure triggered the message and provide the target blood pressure for the patient. The primary care provider will be asked to either evaluate the patient in clinic or manage by telephone. A copy of the message will also be routed to the patient and to the primary oncologist. The investigators will also include a link within the message to an internal Maestro site for further details regarding the blood pressure target levels, a brief description of the chemotherapy the patient is on, and preferred antihypertensive medications in this population. Consistent with the ACC/AHA guidelines for hypertension management, including patients receiving cardiotoxic therapy, the investigators will use the following classification system for the weekly average systolic and diastolic blood pressures. Normal: systolic 95-120 mm Hg, diastolic <80; Elevated: systolic 120-129, diastolic < 80; Stage 1 Hypertension: systolic 130-139, diastolic 80-89; Stage 2 Hypertension: > 140, diastolic > 90. In Phase 2, the investigators will implement and test the clinical pathways and messaging system.

A total of 40 patients with a diagnosis of hypertension who are 18-74 years old who fall under the following criteria will be screened:

* 10 women with Stage 1-III breast cancer who are on active cancer therapy and are receiving either an anthracycline (doxorubicin) or antiHER2 (trastuzumab or pertuzumab)
* 10 men with prostate cancer on androgen deprivation therapy (ADT)
* 10 individuals with CLL on ibrutinib therapy
* 10 HSCT survivors (who had a malignancy)
* Have a smartphone (iPhone or Android)
* Have a Duke primary care provider and Duke oncologist (who is being treated at the Duke Cancer Center)
* Have access or willing to set up access to Duke MyChart (patient portal).
* English speaking patients

The investigators selected these four groups for the following reasons. Stage I-III breast cancer has a 5-year cure rate exceeding 90%. Anthracyclines (doxorubicin) and antiHER2 therapy (trastuzumab or pertuzumab), mainstays of breast cancer therapy, are cardiotoxic and associated with acute and long-term heart failure. Pre-existing hypertension is a key risk factor for development of heart failure in this group. Androgen deprivation therapy is associated with an increased risk of CVD, again, hypertension is a key risk factor for development of CVD in this group. Monotherapy with ibrutinib, or similar novel tyrosine kinase inhibitors, has substantially extended life expectancy for individuals with symptomatic or advanced CLL. Notably, ibrutinib may lead to new onset or progressive hypertension and/or atrial fibrillation. HSCT survivors are exposed to cardiotoxic therapies (anthracyclines, chest radiotherapy) pre-HSCT. Post HSCT complications (GvHD) and chronic comorbidities (hypertension) also contribute to the group's increased risk for developing CVD and congestive heart failure. Thus, blood pressure management is an essential component to improving long-term outcomes for patients in these four groups.

To develop and implement the messaging system, it is important to have the patient, the oncologist, and the primary care provider all in the Duke EHR and patient portal.

ELIGIBILITY:
Inclusion Criteria:

* A total of 40 patients with a diagnosis of hypertension who are 18-74 years old who fall under the following criteria will be screened:

  * 10 women with Stage I-III breast cancer who are on active cancer therapy and are receiving either an anthracycline (doxorubicin) or antiHER2 (trastuzumab or pertuzumab)
  * 10 men with prostate cancer on androgen deprivation therapy (ADT)
  * 10 individuals with CLL on ibrutinib therapy
  * 10 HSCT survivors (who had a malignancy)
  * Have a smartphone (iPhone or Android)
  * Have a Duke primary care provider and Duke oncologist (who is being treated at the Duke Cancer Center)
  * Have access or willing to set up access to Duke MyChart.
  * English speaking patients

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
Patient Adherence | 12 weeks
  To determine the proportions of patients who completed the 3 blood pressure measurements per week (goal of 80% adherence).
Patient Blood Pressure | 12 weeks
  To determine the proportions of patients, by disease group, who have a blood pressure that is above (or below) the target levels.
Primary Care Provider Activation | 12 weeks
  To determine the proportions of primary care providers who (a) received and (b) acted upon the automated message.
End of Study Patient Blood Pressure - Within Target Levels | 1 week (end of study)
  To determine the proportions of patients who are within target levels with the final weekly average pressures.
End of Study Patient Blood Pressure - Outside of Target Levels | 1 week (end of study)
  To determine the proportions of patients who are outside of target levels with the final weekly average pressures.

SECONDARY OUTCOMES:
Clinic-based Blood Pressure | 12 weeks
  To capture all clinic-based blood pressure levels for each patient during the study.
Usability of QardioArm device | 1 week (end of study)
  At the end of the study, a brief REDCap feedback survey of patients to better understand the usability of the QardioArm device will be given.
Acceptability of the Messaging System | 1 week (end of study)
  At the end of the study, a brief REDCap feedback survey of patients and their primary care providers and oncologists to better understand the acceptability of the messaging system and the pathways will be given.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No